CLINICAL TRIAL: NCT00351650
Title: Assessment of Beta Cell Mass in Type 1 Diabetes With 11C-Dihydrotetrabenazine and PET Scan
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060195; 06-DK-0195
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-02-06

CONDITIONS: Type I Diabetes
Keywords: Imaging; Type 1 Diabetes Mellitus (T1DM); Islet; B Cell Mass; Pet Scan; Type 1 Diabetes; T1DM; Pancreas; Healthy Volunteer; HV
MeSH Terms: conditions — Diabetes Mellitus, Type 1

SUMMARY:
This study will test dihydrotetrabenazine, or 11C-DTBZ, a radioactive tracer, as an imaging agent in positron emission tomography (PET). That tracer may have the ability to noninvasively measure beta cell, that is, -cell mass (BCM) in humans. For researchers hoping to develop new treatments for diabetes mellitus, a method of measuring BCM is very important. In this study, researchers will determine if patients with Type 1 diabetes mellitus, who have almost no BCM, have much less pancreatic uptake of the tracer than do patients without diabetes. Patients ages 18 and older may be eligible for this study. Three groups will be studied: Participants who have Type 1 diabetes, those without diabetes, and those who have been successfully treated with a transplant of the pancreas or pancreas and kidney

The study involves three sets of tests that can be done as an outpatient or after being admitted to the hospital. Patients will undergo a medical history and procedures including collection of blood (about 4 teaspoons), pregnancy test for women of childbearing age, magnetic resonance imaging (MRI) scan, PET scan, and tests involving arginine and glucose. Arginine is a substance that stimulates insulin release from the -cells. During the procedure, two intravenous (IV) lines are placed into the arms, one to administer arginine and the other to draw blood (about eight samples during 10 minutes). For the glucose test, patients will drink a solution of dextrose, a sugar, and blood samples will be taken over 2 hours from the IV lines. Some patients experience nausea after drinking the solution. Within 48 hours of either test or both, patients will be placed in the PET scan machine and given an injection of the radioactive material through an IV line. Blood samples of about one-half teaspoon will be drawn before the procedure starts and again every 10 seconds for the first 2 minutes and at several intervals, up to 60 minutes. Finally, patients will also an MRI scan, 30 to 60 minutes long, of the abdomen. This test will be down within two weeks of the PET scan. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. During the scan, patients will be asked to lie still on a table that slides into the tunnel of the scanner. They will be given earplugs, for the machine can be noisy. Patients who have metal within their body that is not compatible with the MRI machine will be withdrawn from the study.

DETAILED DESCRIPTION:
Diabetes is a metabolic disorder in which pancreatic insulin producing B-cells (located in cell clusters called the islets of Langerhans) no longer produce sufficient insulin to maintain an individual's blood sugar concentration within the normal range. Insufficient B-cell function can be caused by an autoimmune killing of the B-cells in type 1 diabetes mellitus (T1DM), or by poorly understood mechanisms in type 2 diabetes mellitus (T2DM). Regardless of the underlying cause, the development of new diabetes treatments is limited by our current inability to objectively measure B-cell mass.

We propose testing a previously used clinical radioligand, dihydrotetrabenazine (DTBZ), as a Positron Emission Tomography (PET) imaging agent for its ability to non-invasively measure B-cell mass in humans. We will study 30 patients, 10 with T1DM, 10 with normal glucose homeostasis, and 5 with a history of T1DM, but successfully restored glucose homeostasis following whole pancreas transplantation. Prior to the PET scans, each patient will undergo metabolic testing to characterize their glucose homeostasis and insulin producing capacity. The pancreas will be initially identified in each patient with high-resolution magnetic resonance imaging (MRI). Then, using anatomical landmarks identified by the MRI, the subject will undergo DTBZ-PET imaging. We predict that the radioactivity signal in the pancreas from the DTBZ-PET images will be significantly different between control subjects and T1DM subjects. Further, we predict that the DTBZ-PET images obtained in individuals with functioning pancreas allografts (and such patients have two pancreases- their native pancreas and their pancreas allografts) will reveal signal intensities from the two glands that correlates closely with each gland's insulin producing capacity. Should these studies suggest DTBZ has merit as a beta cell imaging agent, we will expand the study to include patients with T2DM.

ELIGIBILITY:
* INCLUSION CRITERIA

Patients with T1DM inclusion criteria:

1. Age greater than 18
2. History consistent with T1DM

   1. non-obese (BMI less than 35 kg/m(2)), and
   2. normal insulin sensitivity (as judged by insulin requirements less than or equal to 0.8 unit/kg/day).
   3. Low C-Peptide (less than or equal to 0.6 ng/ml)

Pancreas Transplant Patient inclusion criteria:

1. Age greater than 18
2. History consistent with T1DM (as above) PRIOR to pancreas transplant.
3. Normal pancreas allograft function for at least the preceding 1 year.
4. No acute rejection episodes within the past year.

Control Patient inclusion criteria:

1. Age greater than 18
2. No history of diabetes.
3. Fasting blood glucose less than 100 mg/dl.
4. Normal oral glucose tolerance.
5. BMI less than 35 kg/m(2)

Exclusion criteria for all:

1. Liver dysfunction as determined by history, physical examination, and standard liver function testing (abnormal values for AST, ALT, Total/Direct Bilirubin, Alkaline Phosphatase)
2. Coagulopathy
3. Pregnancy
4. Current breast feeding
5. Use of MAO inhibitors or Levodopa
6. Patients with a contraindication to MRI scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-07-09; Study Completion 2008-02-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Malaisse WJ, Ladriere L, Sener A. Pancreatic fate of 6-deoxy-6-[125I]iodo-D-glucose: in vitro experiments. Endocrine. 2000 Dec;13(3):411-6. PMID 11216655